CLINICAL TRIAL: NCT02408978
Title: Pilot Study of OXP005 to Assess Gastroduodenal Irritation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oxford Pharmascience Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: OXP005-002
Record Dates: First submitted 2015-03-31; First posted 2015-04-06 (Estimated); Last update posted 2015-06-18 (Estimated); Status verified 2015-06

CONDITIONS: Gastroduodenal Erosions
MeSH Terms: interventions — Naproxen

ARMS (2):
- OXP005 (Experimental): 1g naproxen
  Interventions: Drug: OXP005
- naproxen (Active Comparator): 1g naproxen
  Interventions: Drug: Naproxen

INTERVENTIONS:
Drug: OXP005
  Arms: OXP005
Drug: Naproxen
  Arms: naproxen

SUMMARY:
Oxford Pharmascience Ltd (the Sponsor) is developing a new naproxen tablet formulation (the study drug, OXP005), for the potential treatment of rheumatic and painful conditions. The study will compare the study drug to an already marketed formulation of prescription strength naproxen (Naprosyn® the reference product) by looking at the relative impact of both products on gastroduodenal (GD) irritation by performing a specialist procedure called an endoscopy (or more specifically, a gastroscopy). The safety and tolerability of the study drug will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subject
* Healthy, normal upper GI tract as indicated by no ulcers or erosions at baseline, as assessed by the gastroenterologist conducting the endoscopy (ie Lanza score of 0 in both the stomach and duodenum)
* H. pylori negative

Exclusion Criteria:

* Clinically significant abnormal laboratory parameters
* Any clinically significant diseases or conditions affecting the haematopoietic, cardiovascular, renal, hepatic, endocrine, pulmonary, centralcnervous, immunological, dermatological, GI or any other body system

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2015-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Severity of GD irritation in the stomach and duodenum as measured by the Lanza score | Day 8
Total number of GD erosions overall | Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Mair, MBChB, DRCOG, Principal Investigator — Quotient Clinical Ltd
Locations (1):
- Quotient Clinical Ltd, Nottingham, United Kingdom